CLINICAL TRIAL: NCT05227287
Title: Autosomal Dominant Hypocalcemia Types 1 And 2 (ADH1/2) Disease Monitoring Study (DMS)
Brief Title: ADH1 and ADH2 Disease Monitoring Study (DMS)
Acronym: CLARIFY
Status: Active, not recruiting | Type: Observational
Sponsor: Calcilytix Therapeutics, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Other Study IDs: CLTX-305-901
Record Dates: First submitted 2022-01-18; First posted 2022-02-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-08

CONDITIONS: Autosomal Dominant Hypocalcemia
Keywords: Autosomal Dominant Hypocalcemia Type 1 (ADH1); Autosomal Dominant Hypocalcemia Type 2 (ADH2); Hypocalcemia; Musculoskeletal Diseases; Muscular Diseases; Musculoskeletal Abnormalities; Calcium Metabolism Disorders; Metabolic Diseases; Hypoparathyroidism; Hypocalcemic Seizures; Hypercalciuria; Nephrocalcinosis; Nephrolithiasis; Calcium Sensing Receptor; CaSR gene; CaSR gene mutation; CaSR mutation; GNA11 gene; GNA11 gene mutation; GNA11 mutation
MeSH Terms: conditions — Hypercalciuric Hypocalcemia, Familial; Hypocalcemia; Musculoskeletal Diseases; Muscular Diseases; Musculoskeletal Abnormalities; Calcium Metabolism Disorders; Metabolic Diseases; Hypoparathyroidism; Hypercalciuria; Nephrocalcinosis; Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADH 1/2 DMS: Participants with ADH1 or ADH2. No investigational product will be administered to participants in this study. Participants will only receive standard of care (SoC) treatment as directed by the participants' treating physicians.

SUMMARY:
A global, multi-center, Disease Monitoring Study (DMS) in participants with Autosomal Dominant Hypocalcemia Type 1 (ADH1) or Autosomal Dominant Hypocalcemia Type 2 (ADH2) designed to characterize ADH1 and ADH2 disease presentation and progression through retrospective (past) and longitudinal prospective (over time into the future) data collection.

DETAILED DESCRIPTION:
The ADH1 and ADH2 DMS is designed to better understand the disease burden of ADH1 and ADH2, how participants with ADH1 or ADH2 are managed with standard of care practices in a real-world setting, and how standard of care treatment impacts ADH1 and ADH2 symptoms.

The study will include adult and pediatric participants with a confirmed clinical diagnosis of ADH1 or ADH2. Each participant's data will be collected over a period of up to 5 years. In addition, retrospective (or past) data will be collected.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a documented activating variant or variant of uncertain significance of the CASR gene causative of ADH1 or documented activating variant or variant of uncertain significance of the GNA11 gene causative of ADH2 associated with a clinical syndrome of hypoparathyroidism prior to enrollment

Note: Acceptable documentation includes CASR or GNA11 genetic analysis report. If no prior documented CASR or GNA11 gene variant or variant of uncertain significance, potential participants can undergo CASR and GNA11 gene variant analysis at Screening.

* Be willing and able to provide informed consent or assent after the nature of the study and its details have been explained, and prior to any research-related procedures
* Be willing and able to provide access to prior medical records including imaging, biochemical, and diagnostic and medical history data, if available
* Be willing and able to comply with the study visit schedule and study procedures

Key Exclusion Criteria:

* Have serious medical or psychiatric comorbidity that, in the opinion of the Investigator, would present a concern for participant safety or compromise the ability to provide consent or assent, or comply with the study visit schedule and study procedures
* Enrollment in an interventional clinical study at the time of DMS Screening visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants include children (birth to 17 years) and adults (18 - 90 years) with ADH1 or ADH2 as determined by an activating variant of CASR in ADH1 or GNA11 in ADH2.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Blood Calcium Homeostasis | Up to 60 months
Phosphorus Homeostasis | Up to 60 months
Magnesium Homeostasis | Up to 60 months
Intact Parathyroid Hormone (iPTH) Homeostasis | Up to 60 months
Mineral Homeostasis as Assessed by 1,25-dihydroxyvitamin D Homeostasis | Up to 60 months
Urine Calcium Homeostasis | Up to 60 months
Urine Phosphorus Homeostasis | Up to 60 months
Urine Magnesium Homeostasis | Up to 60 months

SECONDARY OUTCOMES:
Blood Creatinine Levels | Up to 60 months
Estimated Glomerular Filtration Rate (eGFR) | Up to 60 months
Number of Participants With Nephrocalcinosis and Nephrolithiasis as Assessed by Renal Ultrasound | Up to 60 months
Bone Mineral Density as Assessed by Dual-Energy X-Ray Absorptiometry (DXA) | Up to 60 months
Change from Baseline in 36-Item Short Form Health Survey (SF-36v2) Physical Component Score and Mental Component Score in Participants ≥ 16 years | Up to 60 months
Change from Baseline in 10-Item Short-Form 10 Healthy Survey for Children (SF-10) Score in participants ≥ 6 years and <16 years | Up to 60 months
Number of Participants Receiving One or More ADH1/2 Treatment Regimens | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Calcilytix Medical Director, Study Director — Calcilytix Therapeutics, Inc., a BridgeBio company
Locations (27):
- United States (9):
  - University of California, San Francisco (UCSF) - Benioff Children's Hospital - Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Indiana University (IU) School of Medicine - University Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Physician's East Endocrinology, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University Medical Center (OSUMC), Columbus, Ohio
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia
- Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant, Belgium
- Bone Research and Education Centre, Oakville, Ontario, Canada
- Aarhus University Hospital, Aarhus, Denmark
- Helsinki University Hospital (HUS) - The New Children's Hospital, Helsinki, Finland
- France (4):
  - HCL Hopital Femme Mere Enfant, Bron, Auvergne-Rhône-Alpes
  - HCL Hopital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes
  - CHU de Lille, Lille
  - Departement d'Endocrinologie et Diabetes pour Enfants - AP-HP Hopital Bicetre, Le Kremlin-Bicêtre, Île-de-France Region
- Endokrinologikum Gottingen, Göttingen, Germany
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Policlinico Universitario Campus Bio-Medico, Rome
- Japan (2):
  - Osaka University Hospital, Osaka
  - The University of Tokyo Hospital, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- Centro Hospitalar Universitario de Lisboa Norte - Hospital de Santa Maria, Lisbon, Portugal
- Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No